CLINICAL TRIAL: NCT03384784
Title: Targeting the Cholinergic Pathway in HIV-associated Inflammation and Cognitive Dysfunction
Brief Title: Effect of Galantamine on Inflammation and Cognition
Acronym: CHI
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 828125; R01DA044906 (NIH)
Record Dates: First submitted 2017-12-08; First posted 2017-12-27 (Actual); Results first posted 2024-10-17 (Actual); Last update posted 2024-10-17 (Actual); Status verified 2024-10

CONDITIONS: HIV Associated Cognitive Motor Complex
Keywords: HIV; Neurocognition; Inflammation; Galantamine; Nicotine; Tobacco Use
MeSH Terms: conditions — AIDS Dementia Complex; Inflammation; Tobacco Use | interventions — Galantamine; Sugars

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Galantamine first (Experimental): This is a crossover study such that all participants receive both placebo and galantamine. Participants were randomized to receive galantamine first and placebo second. Timepoints Week 0 through Week 12 represent the first period and Weeks 16 through 28 represent the second period.
  This study follows the FDA-recommended dosing regimen for galantamine extended release (GAL ER): 4 weeks at 8 mg (once a day), 4 weeks at 16 mg (once a day), and 4 weeks at 24 mg (once a day).
  The University of Pennsylvania Investigational Drug Service (IDS) will oversee the randomization of all study medication, purchase study medication, manufacture matched placebo, encapsulate and package them in blister packs to maintain double-blind procedures.
  Interventions: Drug: Galantamine; Drug: Placebo
- Placebo first (Placebo Comparator): This is a crossover study such that all participants receive both placebo and galantamine. Participants were randomized to receive galantamine first and placebo second. Timepoints Week 0 through Week 12 represent the first period and Weeks 16 through 28 represent the second period.
  Placebo ingredients will be purchased, encapsulated, and packaged into blister packs by the IDS at the University of Pennsylvania. Both active medication and placebo will look identical.
  The study medication assignments for each participant in this project is randomized and counterbalanced. This means that approximately 50% of participants will take galantamine during the first medication period, followed by the placebo in the second medication period. Alternatively, approximately 50% of participants will take the placebo during the first medication period, followed by galantamine during the second medication period.
  Interventions: Drug: Galantamine; Drug: Placebo

INTERVENTIONS:
Drug: Galantamine — The study will be performed using the 8mg, 16mg and 24mg doses of galantamine hydrobromide-ER. The dosing regimen will be an initial 4 weeks of drug run-up at the lowest 8mg q.d. dose, followed by 16mg q.d. for the following 4 weeks, and the dose will be increased for the last 4 weeks to 24mg. Participants will be instructed to take one 8mg 16mg or 24mg pill (galantamine-ER or placebo) every morning, preferably with food.
  Other Names: Razadyne ER
Drug: Placebo — Matched placebo will be made in-house using lactulose filler in gel capsules. Participants will be instructed to take one pills every morning for 12 weeks.
  Other Names: Sugar Pill

SUMMARY:
This study tests whether galantamine (GAL) reduces HIV-related inflammation and cognitive deficits. In this double-blind placebo-controlled crossover study, HIV-infected individuals (N=120; 60 smokers and 60 non-smokers) will be randomized to 12 weeks of GAL or placebo, followed by a 4-week washout, then 12 weeks of GAL or placebo (arms switched). Outcomes are monocyte/macrophage and T cell activation and neurocognitive performance.

DETAILED DESCRIPTION:
Although anti-retroviral therapy (ART) enhances life expectancy and overall quality of life (QoL), HIV-infected individuals are increasingly vulnerable to non-AIDS-related diseases including HIV-associated neurocognitive disorders (HAND). Inflammation is a primary mechanism in the pathogenesis of HAND and tobacco use may further exacerbate inflammation. Conversely, nicotine alone has anti-inflammatory effects suggesting that stimulating the cholinergic pathway via pharmacological treatment [e.g., galantamine (GAL)] may suppress inflammation and reverse or prevent neurocognitive deficits in HIV-1 infection. In this double-blind, placebo-controlled crossover study, HIV-infected individuals (N=120; 60 smokers, 60 nonsmokers) will be randomized to 12 weeks of GAL or placebo, followed by a 4-week washout, then 12 weeks of GAL or placebo (arms switched). All subjects will be stable on ART and the GAL dose will follow FDA guidelines. At the beginning and end of each treatment phase, inflammatory biomarkers and viral load will be assessed. Monocyte transcriptomics will also be assessed on a subset of the sample (n=60; 30/group). Neurocognition and clinical outcomes (e.g., QoL) will be measured at baseline and at 4-week intervals during each treatment phase. The primary outcomes are monocyte/macrophage and T-cell activation (CD16, CD163, and CC chemokine receptor type 2 or CCR2 expression; plasma CC chemokine ligand type 2 or CCL2 [MCP-1 or monocyte chemoattractant protein-1], sCD14; CD38/HLA-DR [cluster of differentiation 38/Human Leukocyte Antigen- antigen D Related] on CD8 [cluster of differentiation 8] cells) and neurocognitive performance (processing speed, verbal learning/memory, executive function). Exploratory outcomes include monocyte gene expression patterns and broad plasma cytokine analysis. This study will provide insight into the interactions among nAChR activation, HIV immune activation and pathogenesis, and tobacco use and has translational and therapeutic implications that could improve health outcomes among HIV-infected individuals.

ELIGIBILITY:
Inclusion Criteria:

Eligible subjects will be males and females:

1. At least 30 years old
2. Diagnosed with HIV-1 infection
3. On stable ART regimens (no changes to treatment within 4 weeks of Intake visit)
4. Viral load of less than or equal to 200 copies/mL
5. Current cluster of differentiation (CD4) counts greater than 200
6. If current or past diagnosis of bipolar disorder, eligible if:

   1. No psychotic features
   2. Montgomery-Asberg Depression Rating Scale (MADRS): total score less than 8 (past 4 weeks), suicidal item score less than 1 (past 4 weeks)
   3. Young Mania Rating Scale (Y-MRS): total score less than 8 (past 4 weeks), irritability, speech content, disruptive or aggressive behavior items score less than 3 (past 4 weeks)
   4. No psychiatric hospitalization or Emergency Room visits for psychiatric issues in the past 6 months
   5. No aggressive or violent acts or behavior in the past 6 months
7. Able to communicate in English and provide written informed consent
8. Will be residing in the geographic area for at least 7 months
9. Not currently trying to quit smoking
10. Smoking Status

    1. Smokers (HIV+S) will report at least 5 instances of smoking per day, on average for the past year and provide a breath carbon monoxide (CO) sample greater than 5 ppm at Intake and at the beginning of each treatment period
    2. Non-smokers (HIV+NS) will report smoking fewer than 100 cigarettes in their lifetime, or less than 5 pack years of smoking and no cigarettes in the last year. They will self-report no current use of any tobacco or nicotine product and will provide a CO sample of less than 3 ppm at Intake and at the beginning of each treatment period. If CO sample does not reflect self-report, the PI will be consulted to determine eligibility.

Exclusion Criteria:

Subjects who present with and/or self-report the following criteria will not be eligible to participate in the study.

Smoking Behavior

1. Current enrollment or plans to enroll in another smoking cessation program in the next 7 months.
2. Regular (daily) use of electronic cigarettes, chewing tobacco, snuff, snus, cigars, cigarillos, or pipes.
3. Current use or plans to use nicotine substitutes (gum, patch, lozenge, e-cigarette) or smoking cessation treatments in the next 7 months.

Alcohol/Drug Use

1. Current untreated and unstable diagnosis of substance abuse or dependence (if past use and if receiving treatment and stable for at least 30 days, eligible)
2. Positive urine drug screen for cocaine, methamphetamines, phencyclidine (PCP), barbiturates, ecstasy (MDMA), at Intake or Lab visits. Those who screen positive for amphetamines, benzodiazepines, methadone, oxycodone, and/or opiates (low level cut-off 300 ng/mL) and who are prescribed these medications will be reviewed on a case-by-case basis by the study physician and PIs (see Measures and Table 1 for details). Participants believed to have a false-positive result on the drug screen may continue in the study, with investigator approval.

Medical/Psychiatric Conditions

1. Women who are pregnant, planning a pregnancy or lactating
2. Current diagnosis of unstable and untreated major depression (if stable for at least 30 days, eligible)
3. Current or past diagnosis of psychotic disorder
4. Cancer diagnosis within the past 6 months (except basal cell carcinoma)
5. Major heart disease or stroke within the past 6 months
6. Uncontrolled hypertension (systolic blood pressure greater than 160 or diastolic blood pressure greater than 100).
7. Medical conditions contraindicated for use with galantamine:

   1. Diagnosis of Alzheimer's disease or dementia
   2. Epilepsy or other seizure disorder
8. Bladder outflow obstruction
9. Active HCV co-infection (if cured, requires study physician approval)
10. Liver function tests more than 20% outside of the normal range; Gamma-glutamyl transpeptidase (GGT) values more than 20% outside of the normal range. If Albumin/Globulin ratios are 20% outside of normal range the abnormal value will be evaluated for clinical significance by the Study Physician and eligibility will determined on a case-by-case basis.
11. Renal disease or renal dysfunction (e.g., serum creatinine levels greater than 1.5 X upper limit of normal). Those with moderate hepatic impairment or creatinine clearance 9 to 59 mL/min shall not exceed the 16 mg/day dose.
12. Peptic ulcer disease (requires study physician approval)
13. Suicide risk as indicated by at least one of the following on the Columbia Suicide Severity Rating Scale (the PI and/or study psychologist will be consulted to assess safety and determine eligibility in cases close to the eligibility cutoffs):

    1. Current suicidal ideation (within 30 days of enrollment)
    2. Two or more lifetime suicide attempts or episodes of suicidal behavior
    3. Any suicide attempt or suicidal behavior within 2 years of enrollment

Medication

1. Current use or discontinuation within the last 14 days of:

   1. Quit smoking medications including varenicline (Chantix), bupropion (Wellbutrin)
   2. Anti-psychotic medications (e.g., Zyprexa, Clozaril, Seroquel, Risperdal). If used to treat psychotic symptoms. Other uses may be eligible pending physician approval).
   3. Systemic Steroids (e.g., Prednisone).
   4. Alzheimer's disease medications (e.g., Acetylcholinesterase inhibitors (ACIs), Aricept/donepezil, Exelon/rivastigmine, Tacrine, or memantine)
   5. Irritable bowel syndrome medication (e.g., Dicyclomine/Bentyl)
   6. Heart medications (e.g., quinidine).
   7. Muscle relaxants (e.g., Anectine/succinylcholine)
   8. Anti-seizure medications (e.g. Ativan, Banzel, Carbatrol, Dilantin, Lamictal, Gabitril, Lyrica, Neurontin, Tegretol, Topomax) if used to treat a seizure disorder or epilepsy. Other uses may be eligible.
   9. Urinary retention medications (e.g., Duvoid/bethanechol, Proscar/finasteride, Avodart/dutasteride, Dibenzyline/ phenoxybenzamine, Regitine/phentolamine)
2. Daily use of:

   1. Opiate-containing medications for chronic pain (Duragesic/fentanyl patches, Percocet, Oxycontin). Smokers who report taking opiate-containing medications on an "as-needed" basis will be instructed to refrain from use until their study participation is over and that they will be tested to ensure they have complied with this requirement.
   2. Chronic obstructive pulmonary disease (COPD) medication (e.g., Atrovent/Ipratropium Bromide)
3. Known allergy to study medication.

Subjects will be instructed to refrain from using any study prohibited drugs/medications (both recreational and prescription) throughout their participation in the study.

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2017-10-30 (Actual); Primary Completion 2022-05-31 (Actual); Study Completion 2022-05-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca L Ashare, PhD, Principal Investigator — University of Pennsylvania
Locations (1):
- Center for Interdisciplinary Research on Nicotine Addiction, University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
The final dataset will include demographic and behavioral assessments and laboratory data bio-specimens. Because the dataset will contain personal health information, identifying information will be collected. Even though the final dataset will be stripped of identifiers prior to release for sharing, investigators will do the following to reduce the possibility confidentiality loss. We will make the data and associated documentation available to users only under a data-sharing agreement that provides for: (1) a commitment to using data only for research purposes and not to identify any individual participant; (2) a commitment to securing the data using appropriate computer technology; and (3) a commitment to destroying or returning the data after analyses are completed.
  Transcriptomic data will be deposited with a public access database such as NCBI's Gene Expression Omnibus (GEO) database (http://www.ncbi.nlm.nih.gov/geo/)
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will be made available starting 6 months after the summary data are published or January 2024 (whichever comes first) and will be made available for 5 years.
Access Criteria: The PIs will review requests for data and all users must sign a data sharing agreement as described above.

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Because there was a gap between enrollment and assignment to group, some participants were lost to follow-up between those time points.
Groups:
- Galantamine First: This is a crossover study such that all participants receive both placebo and galantamine. Participants were randomized to receive galantamine first and placebo second. Timepoints Week 0 through Week 12 represent the first period and Weeks 16 through 28 represent the second period.
  This study follows the FDA-recommended dosing regimen for galantamine extended release (GAL ER): 4 weeks at 8 mg (once a day), 4 weeks at 16 mg (once a day), and 4 weeks at 24 mg (once a day).
  The University of Pennsylvania Investigational Drug Service (IDS) will oversee the randomization of all study medication, purchase study medication, manufacture matched placebo, encapsulate and package them in blister packs to maintain double-blind procedures.
  Galantamine: The study will be performed using the 8mg, 16mg and 24mg doses of galantamine hydrobromide-ER. The dosing regimen will be an initial 4 weeks of drug run-up at the lowest 8mg q.d. dose, followed by 16mg q.d. for the following 4 weeks, and the dose will be increased for the last 4 weeks to 24mg. Participants will be instructed to take one 8mg 16mg or 24mg pill (galantamine-ER or placebo) every morning, preferably with food.
- Placebo First: This is a crossover study such that all participants receive both placebo and galantamine. Participants were randomized to receive placebo first and galantamine second. Timepoints Week 0 through Week 12 represent the first period and Weeks 16 through 28 represent the second period.
  Placebo ingredients will be purchased, encapsulated, and packaged into blister packs by the IDS at the University of Pennsylvania. Both active medication and placebo will look identical.
  The study medication assignments for each participant in this project is randomized and counterbalanced. This means that approximately 50% of participants will take galantamine during the first medication period, followed by the placebo in the second medication period. Alternatively, approximately 50% of participants will take the placebo during the first medication period, followed by galantamine during the second medication period.
  Placebo: Matched placebo will be made in-house using lactulose filler in gel capsules. Participants will be instructed to take one pills every morning for 12 weeks.
Period: First Intervention (12 Weeks)
Arm/Group | Galantamine First | Placebo First
Started | 28 | 30
Completed | 25 | 25
Not Completed | 3 | 5
Period: Washout (4 Weeks)
Arm/Group | Galantamine First | Placebo First
Started | 25 | 25
Completed | 17 | 24
Not Completed | 8 | 1
Period: Second Intervention (12 Weeks)
Arm/Group | Galantamine First | Placebo First
Started | 17 | 24
Completed | 16 | 21
Not Completed | 1 | 3

BASELINE CHARACTERISTICS:
Groups:
- Placebo First: This is a crossover study such that all participants receive both placebo and galantamine. Participants were randomized to receive galantamine first and placebo second. Timepoints Week 0 through Week 12 represent the first period and Weeks 16 through 28 represent the second period.
  Placebo ingredients will be purchased, encapsulated, and packaged into blister packs by the IDS at the University of Pennsylvania. Both active medication and placebo will look identical.
  The study medication assignments for each participant in this project is randomized and counterbalanced. This means that approximately 50% of participants will take galantamine during the first medication period, followed by the placebo in the second medication period. Alternatively, approximately 50% of participants will take the placebo during the first medication period, followed by galantamine during the second medication period.
  Placebo: Matched placebo will be made in-house using lactulose filler in gel capsules. Participants will be instructed to take one pills every morning for 12 weeks.
- Total: Total of all reporting groups
Arm/Group | Galantamine First | Placebo First | Total
Number analyzed (Participants) | 28 | 30 | 58
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 28 | 30 | 58
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.9 (3.7) | 57.3 (5.1) | 57.6 (4.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 8 | 13
  Male | 23 | 22 | 45
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 1 | 4
  Not Hispanic or Latino | 25 | 29 | 54
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 21 | 19 | 40
  White | 4 | 10 | 14
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 2 | 1 | 3
Region of Enrollment [Number; unit: participants]
  United States | 28 | 30 | 58
Smoking History [Count of Participants; unit: Participants]
  Non-Smoker | 10 | 22 | 32
  Current Smoker | 18 | 8 | 26
CD4 Levels at Intake [Mean (Standard Deviation); unit: cells/microliter] | 769.8 (311.2) | 611.6 (201.1) | 687.9 (269.7)
Viral Load at Intake [Count of Participants; unit: Participants]
  Viral load < 50 copies/mL | 25 | 28 | 53
  Viral load > = 50 copies/mL | 3 | 2 | 5

OUTCOME MEASURES:

1. Primary Outcome: Change in Cognition
Description: Cognitive function will be assessed 4 times at Lab Visits. Executive function was measured by the task switch cost from the Color shape task, measured in ms. Executive function was also measured via response time (ms) and accuracy (# correct) on an N-back working memory task. Verbal learning and memory were measured by the Total Recall and Delayed Recall, respectively, from the Hopkins Verbal Learning Test. Response inhibition was measured by the stop signal reaction time (ms) from the Stop Signal Task. A composite score will be created by computed standardized z-scores for each measure (where the mean is 0 and the standard deviation is 1) and then averaging the z-scores. Measures of response time were reverse coded such that higher z-scores indicate better cognitive performance. The primary outcome is the change from baseline cognitive function after 12 weeks of treatment. Change in cognition will be measured during each treatment arm.
Time Frame: Period1 Lab 1 (Week 0), Period 1 Lab 2 (Week 12), Period 2 Lab 1 (Week 16), Period 2 Lab 2 (Week 28)
Population: Number analyzed at each time point reflects participants who had complete data for all cognitive measures.
Measure: Mean (Standard Deviation); unit: Z-score
Arm/Group | Galantamine First | Placebo First
Number analyzed (Participants) | 28 | 30
Z-score
  Period1 Lab 1 (Week 0) | .018 (.469) | .12 (.509)
  Period 1 Lab 2 (Week 12): number analyzed (Participants) | 17 | 20
  Period 1 Lab 2 (Week 12) | 0.068 (0.695) | 0.201 (0.615)
  Period 2 Lab 1 (Week 16): number analyzed (Participants) | 11 | 18
  Period 2 Lab 1 (Week 16) | 0.020 (0.746) | 0.440 (0.578)
  Period 2 Lab 2 (Week 28): number analyzed (Participants) | 11 | 15
  Period 2 Lab 2 (Week 28) | 0.219 (0.806) | 0.490 (0.472)

2. Primary Outcome: Change in Inflammation (MCP-1)
Description: Cellular markers of immune activation will be measured in whole blood and soluble markers of immune activation will be measured in plasma at Lab Visits. The primary outcome is the change in monocyte and T cell surface activation and soluble markers after 12 weeks of treatment. Because this is a within-subject crossover study, changes in cellular markers will be measured during each treatment arm.
Time Frame: Period1 Lab 1 (Week 0), Period 1 Lab 2 (Week 12), Period 2 Lab 1 (Week 16), Period 2 Lab 2 (Week 28)
Population: Number analyzed reflects participants who had complete data at each time point.
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Galantamine First | Placebo First
Number analyzed (Participants) | 28 | 30
pg/mL
  Period1 Lab 1 (Week 0) | 405.00 (277.68) | 402.05 (206.56)
  Period1 Lab 2 (Week 12): number analyzed (Participants) | 19 | 24
  Period1 Lab 2 (Week 12) | 423.33 (266.71) | 337.01 (163.38)
  Period2 Lab 1 (Week 16): number analyzed (Participants) | 17 | 23
  Period2 Lab 1 (Week 16) | 411.71 (221.34) | 350.00 (149.55)
  Period2 Lab 2 (Week 28): number analyzed (Participants) | 14 | 19
  Period2 Lab 2 (Week 28) | 410.76 (300.29) | 334.91 (155.85)

3. Primary Outcome: Change in Inflammation (Percentage of CD14+ Monocytes Expressing CD8)
Description: as for outcome 2
Time Frame: Period1 Lab 1 (Week 0), Period 1 Lab 2 (Week 12), Period 2 Lab 1 (Week 16), Period 2 Lab 2 (Week 28)
Population: Number analyzed reflects participants with complete data for this measure at each time point.
Measure: Mean (Standard Deviation); unit: percentage of monocytes expressing CD8
Arm/Group | Galantamine First | Placebo First
Number analyzed (Participants) | 28 | 30
percentage of monocytes expressing CD8
  Period1 Lab 1 (Week 0) | 7.125 (6.859) | 5.590 (4.528)
  Period 1 Lab 2 (Week 12): number analyzed (Participants) | 19 | 24
  Period 1 Lab 2 (Week 12) | 5.747 (5.789) | 5.221 (3.069)
  Period 2 Lab 1 (Week 16): number analyzed (Participants) | 17 | 23
  Period 2 Lab 1 (Week 16) | 4.329 (2.933) | 6.570 (6.738)
  Period 2 Lab 2 (Week 28): number analyzed (Participants) | 14 | 19
  Period 2 Lab 2 (Week 28) | 6.150 (5.257) | 6.916 (4.658)

4. Primary Outcome: Change in Inflammation (CD14)
Description: as for outcome 2
Time Frame: Period1 Lab 1 (Week 0), Period 1 Lab 2 (Week 12), Period 2 Lab 1 (Week 16), Period 2 Lab 2 (Week 28)
Population: Number analyzed reflects participants with complete data for this measure at each time point.
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Galantamine First | Placebo First
Number analyzed (Participants) | 28 | 30
ng/ml
  Period1 Lab 1 (Week 0): number analyzed (Participants) | 27 | 30
  Period1 Lab 1 (Week 0) | 1672.64 (440.69) | 1645.42 (741.79)
  Period 1 Lab 2 (Week 12): number analyzed (Participants) | 18 | 23
  Period 1 Lab 2 (Week 12) | 1807.66 (461.12) | 1512.70 (498.86)
  Period 2 Lab 1 (Week 16): number analyzed (Participants) | 17 | 23
  Period 2 Lab 1 (Week 16) | 1809.55 (330.04) | 1517.90 (515.77)
  Period 2 Lab 2 (Week 28): number analyzed (Participants) | 14 | 19
  Period 2 Lab 2 (Week 28) | 1631.96 (352.70) | 1521.68 (480.99)

5. Primary Outcome: Change in Inflammation (Percentage of CD14+ Monocytes Expressing CD163)
Description: as for outcome 2
Time Frame: Period1 Lab 1 (Week 0), Period 1 Lab 2 (Week 12), Period 2 Lab 1 (Week 16), Period 2 Lab 2 (Week 28)
Population: Number analyzed reflects participants with complete data for this measure at each time point.
Measure: Mean (Standard Deviation); unit: percentage of monocytes expressing CD163
Arm/Group | Galantamine First | Placebo First
Number analyzed (Participants) | 28 | 30
percentage of monocytes expressing CD163
  Period1 Lab 1 (Week 0) | 88.68 (5.48) | 89.11 (6.99)
  Period 1 Lab 2 (Week 12): number analyzed (Participants) | 19 | 24
  Period 1 Lab 2 (Week 12) | 80.03 (20.67) | 83.90 (17.87)
  Period 2 Lab 1 (Week 16): number analyzed (Participants) | 17 | 23
  Period 2 Lab 1 (Week 16) | 86.64 (7.67) | 87.15 (8.95)
  Period 2 Lab 2 (Week 28): number analyzed (Participants) | 14 | 19
  Period 2 Lab 2 (Week 28) | 86.44 (5.06) | 90.94 (5.24)

6. Primary Outcome: Change in Inflammation (Percentage of CD14+ Monocytes Expressing CD16)
Description: as for outcome 2
Time Frame: Period1 Lab 1 (Week 0), Period 1 Lab 2 (Week 12), Period 2 Lab 1 (Week 16), Period 2 Lab 2 (Week 28)
Population: Number analyzed reflects participants with complete data for this measure at each time point.
Measure: Mean (Standard Deviation); unit: percentage of monocytes expressing CD16
Arm/Group | Galantamine First | Placebo First
Number analyzed (Participants) | 28 | 30
percentage of monocytes expressing CD16
  Period1 Lab 1 (Week 0) | 64.18 (19.49) | 64.90 (20.14)
  Period 1 Lab 2 (Week 12): number analyzed (Participants) | 19 | 24
  Period 1 Lab 2 (Week 12) | 67.44 (17.88) | 68.02 (17.79)
  Period 2 Lab 1 (Week 16): number analyzed (Participants) | 17 | 23
  Period 2 Lab 1 (Week 16) | 74.78 (15.27) | 69.04 (17.37)
  Period 2 Lab 2 (Week 28): number analyzed (Participants) | 14 | 19
  Period 2 Lab 2 (Week 28) | 67.83 (13.23) | 59.78 (21.14)

ADVERSE EVENTS:
Time Frame: 28 weeks: From the start of treatment through the end of treatment
Description: The definitions used do not differ. Adverse event reporting was completed using a symptom checklist, listing all expected side effects for the study drug, which was administered at all study visits and included severity rating and description of the symptom. Participants were also given the opportunity to report any events that were not listed on the checklist, provide a severity rating and description.
Groups:
- Galantamine 8mg: This is a crossover study such that all participants receive both placebo and galantamine. Participants were randomized to receive galantamine first and placebo second.
  This study follows the FDA-recommended dosing regimen for galantamine extended release (GAL ER). This group represents when individuals were on the 8 mg dose (whether it was the first or second period).
- Galantamine 16mg: This is a crossover study such that all participants receive both placebo and galantamine. Participants were randomized to receive galantamine first and placebo second.
  This study follows the FDA-recommended dosing regimen for galantamine extended release (GAL ER). This group represents when individuals were on the 16 mg dose (whether it was the first or second period).
- Galantamine 24mg: This is a crossover study such that all participants receive both placebo and galantamine. Participants were randomized to receive galantamine first and placebo second.
  This study follows the FDA-recommended dosing regimen for galantamine extended release (GAL ER). This group represents when individuals were on the 24 mg dose (whether it was the first or second period).
- Placebo: This is a crossover study such that all participants receive both placebo and galantamine. Participants were randomized to receive galantamine first and placebo second.
  This group represents when individuals were taking placebo (at any point in the study).
Arm/Group | Galantamine 8mg | Galantamine 16mg | Galantamine 24mg | Placebo
All-Cause Mortality (participants affected / at risk) | 1/52 | 0/49 | 0/48 | 0/47
Serious Adverse Events (participants affected / at risk) | 1/52 | 0/49 | 2/48 | 2/47
Other Adverse Events (participants affected / at risk) | 2/52 | 4/49 | 2/48 | 3/47
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Galantamine 8mg (N=52) | Galantamine 16mg (N=49) | Galantamine 24mg (N=48) | Placebo (N=47)
Gastrointestinal Bleeding (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Low Hemoglobin (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bone fracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pulled muscle (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Galantamine 8mg (N=52) | Galantamine 16mg (N=49) | Galantamine 24mg (N=48) | Placebo (N=47)
Depression (Psychiatric disorders) | 1 (1) | 2 (2) | 1 (1) | 2 (2)
Fatigue (General disorders) | 1 (1) | 4 (4) | 1 (1) | 1 (4)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-02-22): https://cdn.clinicaltrials.gov/large-docs/84/NCT03384784/Prot_SAP_000.pdf
  • Informed Consent Form (2021-02-22): https://cdn.clinicaltrials.gov/large-docs/84/NCT03384784/ICF_001.pdf